CLINICAL TRIAL: NCT03020303
Title: Aldosterone bloCkade for Health Improvement EValuation in End-stage Renal Disease
Acronym: ACHIEVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACHIEVE Trial
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Endstage Renal Disease
MeSH Terms: interventions — Spironolactone; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Oral Tablet (Placebo Comparator): A tablet with no active medication that will be an exact match of the active spironolactone in taste and appearance
  Interventions: Drug: Placebo Oral Tablet
- Spironolactone 25 MG Tablet (Active Comparator): 25 mg of active spironolactone in tablet form
  Interventions: Drug: Spironolactone 25Mg Tablet

INTERVENTIONS:
Drug: Spironolactone 25Mg Tablet — Randomized participants will receive a study supply of spironolactone 25 mg tablets. They will be instructed to take 1 tablet daily.
  Arms: Spironolactone 25 MG Tablet
Drug: Placebo Oral Tablet — Randomized participants will receive a study supply of placebo tablets with no active medical ingredients. They will be instructed to take 1 tablet daily.
  Arms: Placebo Oral Tablet

SUMMARY:
Individuals receiving dialysis are at risk of heart failure and heart related death. There is an urgent need for treatments that reduce the risk of these problems in patients that require dialysis.

Spironolactone is a pill used to prevent heart failure and related deaths in patients that do not require dialysis. It works by blocking a hormone (aldosterone) in your body that causes high blood pressure and can damage the heart. Although spironolactone is very effective in patients that do not require dialysis, we do not know if spironolactone is effective in dialysis patients. Our research will help determine if spironolactone reduces heart failure and heart related deaths in dialysis patients.

The purpose of this study is to determine if spironolactone reduces death or hospitalization for heart failure and is well tolerated in patients that require dialysis.

DETAILED DESCRIPTION:
Globally, over 2 million people receive dialysis for end-stage renal disease (ESRD) and 650,000 new patients start dialysis each year. Furthermore, the number of patients receiving dialysis is increasing as access to dialysis in the developing world improves and the prevalence of diabetes and vascular disease rises. Despite technical advances in dialysis, the outcomes for patients with ESRD are poor. Patients have frequent hospitalizations, poor health related quality of life and strikingly, high mortality rates.

The most common cause of death in patients receiving dialysis is cardiovascular disease, accounting for >40% of all deaths. Observational studies suggest a causal pathway to cardiovascular death that includes progressive ventricular hypertrophy and dilatation as well as accelerated atherosclerosis. These changes result in myocardial ischemia and cardiac fibrosis that, in turn, lead to heart failure, arrhythmias and cardiac arrest. Strongly implicated in this pathophysiology is aldosterone. Mineralocorticoid receptor antagonists (MRAs) in non-ESRD patients, prevent cardiovascular deaths and small randomized controlled trials of MRAs in ESRD suggests they may reduce death and may be safe.

Spironolactone is the most commonly used MRA worldwide. We will conduct a multicentre randomized controlled trial (RCT) to determine if spironolactone reduces cardiac mortality and hospitalizations for heart failure in patients treated with dialysis. This trial is called the Aldosterone bloCkade for Health Improvement EValuation in End-stage renal disease (ACHIEVE).

ELIGIBILITY:
Inclusion Criteria:

1. Age

   1. ≥45 years or
   2. ≥18 with a history of diabetes
2. On dialysis ≥ 90 days
3. On either

   1. Hemodialysis prescribed at least 2 treatments per week or
   2. Peritoneal dialysis prescribed with at least 1 exchange daily
4. Provides informed consent

Exclusion Criteria:

1. Hyperkalemia

   1. Serum potassium >5.8 mmol/L in the 6 weeks prior to enrollment or
   2. Serum potassium >6.0 mmol/L during active run-in
2. Currently taking and unable to withdraw a mineralocorticoid receptor antagonist (i.e. spironolactone or eplerenone).
3. Known sensitivity or allergy to spironolactone
4. Current or planned pregnancy or breastfeeding
5. Scheduled living related donor renal transplant
6. Life expectancy < 6 months in the opinion of a treating nephrologist.
7. Enrolled in another interventional trial testing a mineralocorticoid receptor antagonist or drug that has a known or likely interaction with spironolactone.
8. Treating physician believes either spironolactone is either absolutely indicated or absolutely contra-indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2538 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
CV Death or Hospitalization for Heart Failure | up to 5 years

SECONDARY OUTCOMES:
Cause specific death | up to 5 years
Hospitalization for Heart Failure | up to 5 years
All-cause death | up to 5 years
All-cause Hospitalization | up to 5 years
Hospitalization for hyperkalemia | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Walsh, MD, PhD, Principal Investigator — McMaster University; PJ Devereaux, MD, PhD, Study Chair — McMaster University
Locations (141):
- Australia (10):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Northern Beaches Hospital, Frenchs Forest, New South Wales
  - Royal North Shore Hospital, Wahroonga, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Health, Clayton, Victoria
  - Western Health - Sunshine Hospital, Saint Albans, Victoria
- Brazil (16):
  - Santa Casa de Misericordia de Belo Horizonte, Santa Efigênia, Belo Horizonte
  - Medical School of Botucatu of the Paulista State University - UNESP, Rubião Júnior, Botucatu
  - Fundacao Pro-Rim, Boa Vista, Joinville
  - Felicio Rocho Foundation - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Fundacao Hospitalar Sao Francisco de Assis, Belo Horizonte, Minas Gerais
  - Servico Ubaense de Nefrologia Ltda, Ubá, Minas Gerais
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul, Paraná
  - Instituto Pro Renal Brazil, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericordia de Porto Alegre -ISCMPA, Bairro Santa Teresa, Porto Alegre
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Arquidiocesano Consul Carlos Reneaux, Brusque, Santa Catarina
  - PROCARDIO Clinica Cardiologica, Blumenau, South Carolina
  - Praxis Pesquisa Medica S/S, Santo André, São Paulo
  - Santa Casa de Misericordia de Votuporanga, Votuporanga, São Paulo
  - Hospital Alemao Oswaldo Cruz, Bela Vista
  - Santa Casa de Misericordia de Ponta Grossa, Ponta Grossa
- Canada (21):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Royal Inland Hospital, Kamloops, British Colombia
  - Kelowna General Hospital, Kelowna, British Colombia
  - St. Pauls Hospital, Vancouver, British Colombia
  - Penticton Regional Hospital, Penticton, British Columbia
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - Cape Breton Regional Hospital, Sydney, Nova Scotia
  - Health Sciences North Research Institute, Greater Sudbury, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Queens University at Kingston General Hospital, Division of Nephrology, Kingston, Ontario
  - Victoria Hospital, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - St. Josephs, Toronto, Toronto, Ontario
  - Humber River Health, Toronto, Ontario
  - CIUSSS Hopital Maisonneuve- Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - The Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec L'Hotel-Dieu de Quebec, Québec, Quebec
- China (24):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - Beijing Miyun District Hospital, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Emergency General Hospital, Beijing
  - Faw General Hospital of Jilin Province, Changchun
  - The Central Hospital of Enshi Tujia and Miao Autonomous Prefecture, Enshi
  - Huai'an First Peoples Hospital, Huai'an
  - The First Hospital of Kunming, Kunming
  - Gansu Baoshihua Hospital, Lanzhou
  - Yichuan County Traditional Chinese Medicine Hospital, Luoyang
  - Shanghai Tongji Hospital, Shanghai
  - Shanxi Provincial Peoples Hospital, Shanxi
  - Shuyang County Hospital of Traditional Chinese Medicine, Suqian
  - Sihong County Fenjinting Hospital, Suqian
  - Tianjin Fifth Central Hospital, Tianjin
  - Tianjin Third Central Hospital, Tianjin
  - Tongiao City Hospital, Tongliao
  - Xinxiang First Peoples Hospital, Xinxiang
  - General Hospital of Xuzhou Mining Group, Xuzhou
  - Peoples Hospital of Yuxi City, Yuxi
  - Peoples Hospital of Zhongwei, Zhongwei
- Ecuador (2):
  - Clinefnorte CIA Ltda, Quito, Pichincha
  - Nefromedic SA, Quito, Pichincha
- India (20):
  - Madras Medical College Chennai, Park Town, Chennai
  - Narayana Hrudayalaya Limited, Bangalore, Karnataka
  - Fortis Hospitals, Bengaluru, Karnataka
  - K S Hegde Medical Academy, Mangaluru, Karnataka
  - Nanjappa Hospitals Shimoga, Shimoga, Karnataka
  - AsterMedCity, Kochi, Kerala
  - Caritas Hospital, Kottayam, Kerala
  - AIMS Hospital Mumbai, Dombivali, Maharashtra
  - National Health and Education Society, Mumbai, Maharashtra
  - Ashirwad Hospital Mumbai, Mumbai, Maharashtra
  - Dhadiwal Hospital, Nashik, Maharashtra
  - ACE Hospital Une, Pune, Maharashtra
  - Aditya Birla Hospital, Pune, Maharashtra
  - Vijaya Hospital, Chennai, Tamil Nadu
  - Apollo Hospitals, Chennai, Tamil Nadu
  - Nizams Institute of Medical Sciences, Hyderabad, Telangana
  - Osmania General Hospital, Hyderabad, Telegana
  - Government Rajaji Hospital, Madurai, Madurai
  - Father Muller Medical College, Mangalore
  - Seven Star Hospital, Nagpur
- Malaysia (12):
  - Hospital Sultanah Aminah, Johor Bahru, Johor Bahru, Johor
  - Hospital Pakar Sultanah Fatimah, Muar town, Johor
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre (UMMC), Kuala Lumpur, Kuala Lumpur
  - Hospital Sultanah Nur Zahirah Kuala Terengganu, Kuala Terengganu, Kuala Terengganu
  - Hospital Taiping, Taiping, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Kajang, Kajang, Selangor
  - Hospital Tengku Ampuan Rahimah Klang, Klang, Selangor
  - Hospital Tengku Ampuan Afzan, Kuantan, Kuantan
  - Hospital Tuanku Jaafar, Seremban, Seremban
  - Hospital Ampang, Setapak
- New Zealand (6):
  - North Shore Hospital, Takapuna, Auckland
  - Waikato Hospital, Hamilton, Waikato Region
  - Dunedin Hospital, Dunedin
  - Hawkes Bay Hospital, Hastings
  - Palmerston North Hospital, Palmerston North
  - Whangarei Hospital, Whangarei
- Philippines (2):
  - Philippines General Hospital, Ermita, Manila
  - National Kidney and Transplant Institute, Quezon City, Manila
- Turkey (Türkiye) (3):
  - Hacettepe University Hospitals Hemodialysis Center, Ankara
  - Osmangazi University, Eskişehir
  - Memorial Service Hospital, Istanbul
- United Kingdom (21):
  - Ulster Hospital, Dundonald, Belfast
  - Southmead Hospital, Bristol, Bristol
  - University Hospital of Whales Health Park, Cardiff, Cardiff
  - Daisy Hill Hospital, Newry, Down
  - Queen Elizabeth University Hospital, Glasgow, Glasgow
  - East Kent Canterbury Hospital, Canterbury, Kent
  - The Royal London Hospital, London, London
  - Kings College Hospital, London, London
  - City Hospital, Nottingham, Nottingham
  - Churchill Hospital, Headington, Oxford
  - Salford Royal Hospital, Salford, Salford
  - Aberdeen Royal Infirmary, Aberdeen
  - Belfast City Hospital, Belfast
  - Birmingham Hospitals, Birmingham
  - Epsom St. Helier, Carshalton
  - Royal Derby Hospital, Derby
  - Ninewells Hospital, Dundee
  - Leicester General Hospital, Leicester
  - Liverpool University Hospitals, Liverpool
  - South Tees James Cook Hospital, Middlesbrough
  - Royal Stoke University Hospital, Stoke-on-Trent
- Uruguay (4):
  - Canimel Center, Melo, Departamento de Cerro Largo
  - SEDIC Center, Montevideo, Montevideo Department
  - Cedina Center, Montevideo
  - Centro de Asistencia del Sindicato Medico del Uruguay-Institucion de Asistencia medica Privada (CASMU-IAMPP), Montevideo

IPD SHARING:
Plan to Share IPD: No
N/A - no plan to make IPD available to other researchers

REFERENCES:
- [Background] Quach K, Lvtvyn L, Baigent C, Bueti J, Garg AX, Hawley C, Haynes R, Manns B, Perkovic V, Rabbat CG, Wald R, Walsh M. The Safety and Efficacy of Mineralocorticoid Receptor Antagonists in Patients Who Require Dialysis: A Systematic Review and Meta-analysis. Am J Kidney Dis. 2016 Oct;68(4):591-598. doi: 10.1053/j.ajkd.2016.04.011. Epub 2016 Jun 3. PMID 27265777
- [Background] Walsh M, Manns B, Garg AX, Bueti J, Rabbat C, Smyth A, Tyrwhitt J, Bosch J, Gao P, Devereaux PJ, Wald R. The Safety of Eplerenone in Hemodialysis Patients: A Noninferiority Randomized Controlled Trial. Clin J Am Soc Nephrol. 2015 Sep 4;10(9):1602-8. doi: 10.2215/CJN.12371214. Epub 2015 Jul 2. PMID 26138259
- [Derived] Walsh M, Collister D, Gallagher M, Mark PB, de Zoysa JR, Tyrwhitt J, Tennankore K, Reis G, Xavier D, Liu WJ, Zuo L, Wang AY, Felix C, Sola L, Arici M, Villanueva R, Jha V, Precoma D, Rabbat CG, Alavudeen SS, Faruqui AR, Lopez-Flecher M, Pyne L, Wald R, Yuan F, Balasubramanian K, Lee SF, Kuptsova A, Christou C, Devereaux PJ; ACHIEVE Investigators. Spironolactone versus placebo in patients undergoing maintenance dialysis (ACHIEVE): an international, parallel-group, randomised controlled trial. Lancet. 2025 Aug 16;406(10504):695-704. doi: 10.1016/S0140-6736(25)01198-5. PMID 40818850
- [Derived] Walsh M, Collister D, Gallagher M, Mark PB, de Zoysa JR, Tyrwhitt J, Tennankore K, Sola L, Reis G, Xavier D, Villanueva R, Liu WJ, Felix C, Zuo L, Arici M, Jha V, Wald R, Wang AY, Faruqui AR, Yuan F, Lee SF, Kuptsova A, Christou C, Devereaux PJ; ACHIEVE Investigators. The Aldosterone Blockade for Health Improvement Evaluation in End-Stage Renal Disease (ACHIEVE) Trial: Rationale and Clinical Research Protocol. Can J Kidney Health Dis. 2025 Jun 3;12:20543581251348187. doi: 10.1177/20543581251348187. eCollection 2025. PMID 40470466
- [Derived] Huang B, McDowell G, Rao A, Lip GYH. Mineralocorticoid receptor antagonist for chronic kidney disease, risk or benefit? J Hypertens. 2024 Mar 1;42(3):396-398. doi: 10.1097/HJH.0000000000003643. Epub 2024 Feb 1. No abstract available. PMID 38289999
- [Derived] Soomro QH, Charytan DM. Mineralocorticoid Receptor Antagonists and Cardiovascular Health with Kidney Failure. Clin J Am Soc Nephrol. 2021 Jun;16(6):843-845. doi: 10.2215/CJN.04460421. No abstract available. PMID 34117077
- [Derived] Collister D, Mbuagbaw L, Guyatt G, Devereaux PJ, Tennankore KK, Reis G, Sola L, Xavier D, Jha V, Gallagher M, Dans AL, Liu W, de Zoysa J, Felix C, Mark PB, Li Z, Tyrwhitt J, Wilkinson J, Sheridan P, Yuan F, Walsh M; ACHIEVE investigators. Three week compared to seven week run-in period length and the assessment of pre-randomization adherence: A study within a trial. Contemp Clin Trials. 2021 Aug;107:106466. doi: 10.1016/j.cct.2021.106466. Epub 2021 Jun 5. PMID 34098039
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138